CLINICAL TRIAL: NCT05482295
Title: Immunogenicity and Safety Following In-House Recombinant Hepatitis B (Bio Farma) Vaccine Compared to Registered Hepatitis B Vaccine in Indonesian Population (Phase III)
Brief Title: Immunogenicity and Safety Following In-House Recombinant Hepatitis B Vaccine in Indonesian Population (Phase III)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Collaborators: RS Prof. Dr. I.G.N.G Ngoerah (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HepB 0322
Record Dates: First submitted 2022-07-29; First posted 2022-08-01 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Vaccine Reaction; Vaccine Adverse Reaction
Keywords: Hepatitis B vaccine, Vaccine
MeSH Terms: conditions — Hepatitis B | interventions — Vaccines; Engerix-B

STUDY DESIGN:
Intervention Model Description: Experimental, randomized, observer-blind, lot to lot consistency
Who Masked: Participant, Investigator
Masking Description: The subject will be randomized and vaccinated per treatment group by unblinded team.
  The randomization list will be provided by unblinded personel of study team. This unblinded team will keep the list until Bio Farma formally issue the result of the study. Treatment will be allocated in accordance with a randomization list, so that to each randomization number, corresponds only one strictly randomly assigned treatment group (A/B/C/D).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- In-House Recombinant Hepatitis B (Bio Farma) vaccine Batch 1 (Experimental): 3 doses In-House Recombinant Hepatitis B (Bio Farma) vaccine
  Interventions: Biological: In-House Recombinant Hepatitis B (Bio Farma) vaccine
- In-House Recombinant Hepatitis B (Bio Farma) vaccine Batch 2 (Experimental): 3 doses In-House Recombinant Hepatitis B (Bio Farma) vaccine
  Interventions: Biological: In-House Recombinant Hepatitis B (Bio Farma) vaccine
- In-House Recombinant Hepatitis B (Bio Farma) vaccine Batch 3 (Experimental): 3 doses In-House Recombinant Hepatitis B (Bio Farma) vaccine
  Interventions: Biological: In-House Recombinant Hepatitis B (Bio Farma) vaccine
- Registered Hepatitis B vaccine recombinant (Engerix-B) (Active Comparator): 3 doses Registered Hepatitis B vaccine recombinant (Engerix-B)
  Interventions: Biological: Registered Hepatitis B vaccine recombinant (Engerix-B)

INTERVENTIONS:
Biological: In-House Recombinant Hepatitis B (Bio Farma) vaccine — 3 doses of In-House Recombinant Hepatitis B (Bio Farma) vaccine
  Arms: In-House Recombinant Hepatitis B (Bio Farma) vaccine Batch 1; In-House Recombinant Hepatitis B (Bio Farma) vaccine Batch 2; In-House Recombinant Hepatitis B (Bio Farma) vaccine Batch 3
Biological: Registered Hepatitis B vaccine recombinant (Engerix-B) — 3 doses of Registered Hepatitis B vaccine recombinant (Engerix-B)
  Arms: Registered Hepatitis B vaccine recombinant (Engerix-B)

SUMMARY:
This is a phase 3, experimental, randomized, observer-blind, lot to lot consistency study. The primary objective of this study is to assess the protectivity of In-House Recombinant Hepatitis B vaccine 28 days after 3 doses immunization.

DETAILED DESCRIPTION:
This is a phase 3, experimental, randomized, observer-blind, lot to lot consistency study. A total of 540 subjects will be involved in this study.

The primary objective of this study is to assess the protectivity of In-House Recombinant Hepatitis B vaccine 28 days after 3 doses immunization.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individual aged 10 - 50 years old, as determined by clinical judgment, including a medical history and physical exam which confirms the absence of a current or past disease state considered significant by the investigator.
2. Subjects/parents/guardian(s) have been informed properly regarding the study and signed the informed consent form/ informed assent form.
3. Subject/parents/guardian(s) will commit to comply with the instructions of the investigator and the schedule of the trial.

Exclusion Criteria:

1. Subject concomitantly enrolled or scheduled to be enrolled in another trial.
2. Subjects with known history of Hepatitis B contained vaccination in the last 10 years.
3. Evolving severe illness and/or chronic disease and fever (axillary temperature >= 37.5 C) within the 48 hours preceding enrollment.
4. Known history of allergy to any component of the vaccines (based on anamnesis).
5. HBsAg positive.
6. Known history of immunodeficiency disorder (HIV infection, leukemia, lymphoma, or malignancy).
7. History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection.
8. Subject who has received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products or corticosteroid therapy and other immunosuppressant.
9. Pregnancy & Lactation (Adult).
10. Subject already immunized with any vaccine within 4 weeks prior and expects to receive other vaccines within 4 weeks following immunization.

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 540 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Protectivity | 28 days after the primary series of Hepatitis B vaccination
  Number & percentage of subjects with anti HBsAg > 10mIU/ml

SECONDARY OUTCOMES:
Immunogenicity: Serological response | 28 days after the primary series of Hepatitis B vaccination
  Geometric mean of anti-HBsAg, percentage of subjects with increasing antibody titer >= 4 times and/ or percentage of subjects with transition of seronegative to seropositive
Immunogenicity: comparison between IP & control | 28 days after the primary series of Hepatitis B vaccination
  Comparison of GMT, seroprotection, percentage of subjects with increasing antibody titer >=4 times and/ or percentage of subjects with transition of seronegative to seropositive
Immunogenicity: comparison among each batch of IP | 28 days after the primary series of Hepatitis B vaccination
  Comparison of GMT, seroprotection, percentage of subjects with increasing antibody titer >=4 times and/ or percentage of subjects with transition of seronegative to seropositive
Safety: Immediate reaction, Local and systemic events | within the first 30 minutes, after 30 minutes to 7 days, after 7 days to 28 days after each injection
  Immediate reaction, Local and systemic events
Safety: Serious adverse event | from inclusion until 28 days after the last injection
  Any serious adverse event
Safety: Comparison of adverse events between Investigational Products (Hepatitis B) and Control | 28 days after each dose
  Adverse events occuring until 28 days after vaccination
Safety: Comparison of adverse events between each lot number of Recombinant Hepatitis B | 28 days after each dose
  Adverse events occuring until 28 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Trisna Windiani, MD, Principal Investigator — RSUP Prof. dr. I.G.N.G. Ngoerah

IPD SHARING:
Plan to Share IPD: No